CLINICAL TRIAL: NCT02153866
Title: The Safety and Immunogenicity Study of Rotavirus Vaccine Simultaneously Vaccinated With MR or MMR Vaccine
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Sichuan Center for Disease Control and Prevention (Other Government)
Collaborators: China National Biotec Group Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: cnbg-001
Record Dates: First submitted 2014-05-26; First posted 2014-06-03 (Estimated); Last update posted 2014-06-03 (Estimated); Status verified 2014-05

CONDITIONS: Rotavirus
Keywords: rotavirus vaccine
MeSH Terms: interventions — Rotavirus Vaccines; Measles-Mumps-Rubella Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- rotavirus (Placebo Comparator): vaccinate one dose rotavirus vaccine for each of 700 participants aged 8~9months
  Interventions: Biological: rotavirus vaccine
- measles-rubella (Placebo Comparator): vaccinate one dose measles-rubella vaccine for each of 350 participants aged 8~9 months.
  Interventions: Biological: measles-rubella vaccine
- measles-mumps-rubella (Placebo Comparator): vaccinate one dose measles-mumps-rubella vaccine for each of 350 participants aged 8~9 months.
  Interventions: Biological: measles-mumps-rubella vaccine
- rotavirus, measles-rubella (Experimental): simultaneously vaccinate one dose rotavirus vaccine and one dose measles-rubella vaccine for each of 700 participants aged 8~9 months.
  Interventions: Biological: rotavirus vaccine; Biological: measles-rubella vaccine
- rotavirus, measles-mumps-rubella (Experimental): simultaneously vaccinate one dose rotavirus vaccine and one dose measles-mumps-rubella vaccine for each of 700 participants aged 8~9 months.
  Interventions: Biological: rotavirus vaccine; Biological: measles-mumps-rubella vaccine

INTERVENTIONS:
Biological: rotavirus vaccine — 3ml/dose, oral
  Arms: rotavirus; rotavirus, measles-mumps-rubella; rotavirus, measles-rubella
Biological: measles-rubella vaccine — 0.5ml per dose, subcutaneous injection
  Other Names: measles-rubella live attenuated vaccine
  Arms: measles-rubella; rotavirus, measles-rubella
Biological: measles-mumps-rubella vaccine — 0.5ml per dose, subcutaneous injection
  Other Names: measles-mumps-rubella live attenuated vaccine
  Arms: measles-mumps-rubella; rotavirus, measles-mumps-rubella

SUMMARY:
Nowadays these are some vaccines being vaccinated simultaneously, and a doubt is aroused if the safety and immunogenicity are same between inoculating several vaccines simultaneously and inoculating individually. So we carry out this study.

The purpose of this study is to evaluate the difference of safety and immunogenicity on vaccinating rotavirus vaccine simultaneously with measles-rubella vaccine(MR) or measles-mumps-rubella vaccine(MMR) compared to vaccinating rotavirus vaccine, MR or MMR individually.

DETAILED DESCRIPTION:
1. Quality control plan:

   1. All vaccinators should get professional training held by local Health Bureau, and be qualified by local Health Bureau.
   2. All the clinical trial related staffs are trained by provincial or prefectural Center for Disease Control and prevention (CDC) at the beginning.
   3. Provincial and prefectural CDCs conduct supervision at each step, especially during field vaccination and Adverse Events Following Immunization (AEFI) investigation.
   4. Data valid check is designed to work in the database inputting, double entry and validation is also required.
   5. The field works are conduct under SOP (Standard Operating Procedures), The SOP for vaccination procedures which include vaccinee recruitment and vaccination practice etc. is 'Immunization Work Specification' issued by China Ministry of Health in 2005. The SOP for AEFI surveillance is 'AEFI surveillance guideline' issued by China Ministry of Health in 2010.
2. Statistical plan

   1. Safety evaluation The analytic data include all reactions or events within 30 days after vaccination, compare the incidence of reactions among different vaccines, the statistical method is chi-square.
   2. Immunogenicity evaluation Compare the antibody positive rate and Geometric Mean Concentration between pre-vaccination and post-vaccination, and among different vaccine combinations.
3. safety evaluation method

   At the time of vaccination, vaccinees were instructed to report any adverse event to physicians or vaccination providers. Adverse events that were fatal or that resulted in disability and clusters of events (i.e., notably high numbers of similar adverse events related to a certain vaccine) were required to be reported within 2 hours after their occurrence. The following adverse events were required to be reported within 2 days after their occurrence: anaphylaxis or other allergic reactions occurring within 24 hours after vaccination; fever (axillary temperature, >38.5°C), angioedema, or a local injection-site reaction (diameter, >2.5 cm) occurring within 5 days after vaccination; purpura, an Arthus reaction, febrile convulsion, seizure, or polyneuritis occurring within 15 days after vaccination. Other reactions that were common and minor (e.g., mild pain and fatigue) were not required to be reported.
4. Immunogenicity evaluation

Enzyme-linked immunosorbent assay (abbreviated as ELSIA) is used to quantitatively test immunoglobulin G (IgG) of measles, rubella, mumps, test kit is provided by Virion\Serion company. Rotavirus Immunoglobulin A (RV-IgA) is used to test the antibody of rotavirus.

ELIGIBILITY:
Inclusion Criteria:

* Aged 8~9 months healthy child
* Subjects or guardians who can and will comply with the requirements of the protocol
* Without vaccination history of rotavirus vaccine, measles-rubella vaccine and measles-mumps-rubella vaccine.
* Axillary temperature is under 37.0℃.
* Accord with the requirement of drug manual of rotavirus vaccine,measles-rubella vaccine and measles-mumps-rubella vaccine.

Exclusion Criteria:

* Allergic to any component of the vaccines.
* Women of pregnancy, lactation or about to be pregnant in 60 days.
* Infected by some rash disease within one month.
* Known severe immunodeficiency (e.g., from hematologic and solid tumors, receipt of chemotherapy, congenital immunodeficiency, or long-term immunosuppressive therapy or patients with HIV infection who are severely immunocompromised).
* Any prior administration of immunoglobulins, any other vaccines or experimental drugs in the last 4 weeks.
* Family history of seizures or progressive neurological disease.
* Diarrheal caused by rotavirus or lasting for 3 or more days.
* Any condition that in the opinion of the investigator, may interfere with the evaluation of study objectives.

Ages: 8 Months to 9 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2800 (Estimated)
Dates: Start 2013-12; Primary Completion 2014-05 (Actual); Study Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
the occurrence rate of general reaction of different vaccination groups | 1 months after vaccination
  general reaction includes fever (axillary temperature> 3.85℃), local injection-site reaction (diameter> 2.5 cm) etc.

SECONDARY OUTCOMES:
the occurrence rate of severe adverse event of different vaccination groups | 1 month after vaccination
  severe reaction include: anaphylaxis, angioedema, purpura, an Arthus reaction, febrile convulsion, seizure, polyneuritis, other adverse events cause fatal, result in disability or clusters of events (i.e., notably high numbers of similar adverse events related to a certain vaccine)
The variation of antibody Geometric Mean Titer compared between before and after vaccination | 1 month after vaccination
  this measure is used to assess the immunogenicity of different groups

CONTACTS AND LOCATIONS:
Overall Officials: rui ao, Master, Study Director — Sichuan Provincial Center for Disease Control and Prevention